CLINICAL TRIAL: NCT03137602
Title: ATOMIC (Active Teens With MultIple sClerosis) Teens: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Alabama at Birmingham (Other); Queen's University (Other)
Responsible Party: Principal Investigator, E. Ann Yeh, Associate Scientist, Research Institute, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000055499
Record Dates: First submitted 2017-01-03; First posted 2017-05-03 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Pediatric Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATOMIC mobile app (Other): The proposed ATOMIC intervention consists of four primary components: (a) one-on-one chats with a PA coach, (b) informational posts, (c) PA self-monitoring through an activity tracker and (d) educational modules regarding different aspects of becoming PA delivered through our MS specific PA app.
  Interventions: Device: ATOMIC mobile app

INTERVENTIONS:
Device: ATOMIC mobile app — (a) PA Coach, One-on-one Chats. Coaches will conduct three one-on-one phone or video conferencing sessions and will also conduct a text messaging session once per week to reinforce and follow-up on the one-on-one phone sessions during the course of the intervention. (b) PA-Self Monitoring. An activity tracker (Fitbit Charge 2) will be used to allow participants to monitor their activity behaviors (e.g. step counts). (c) PA Information. In addition the coach will send weekly tailored PA informational posts/messages aligned with Social Cognitive Theory (SCT) to all participants. (d) Educational Modules. MS specific web-based interactive PA modules will be provided to patients.

SUMMARY:
Taking part in recommended levels of physical activity in youth with MS may have an important and positive impact on disease symptoms, long-term disability and health outcomes. Unfortunately, youth with MS are highly inactive. In order to address this issue, the investigators have developed an MS-specific mobile application for teens called Active Teens with Multiple Sclerosis (ATOMIC). In this research the investigators will evaluate the feasibility of using the ATOMIC program in youth with MS. The results of this pilot study will provide the data necessary to ensure the ATOMIC program aligns with the needs of youth with MS.

ELIGIBILITY:
Inclusion Criteria:

1. MS diagnosis following standard definitions (IPMSSG);
2. EDSS <4.0;
3. Ability to speak English.

Exclusion Criteria:

1. Known cardiac disease, including cyanotic congenital heart disease;
2. inability to understand instructions and tolerate proposed testing or vigorous PA.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the ATOMIC program | Entire study - up to 24 weeks
  Determined by calculating accrual rates, drop-out rates, adherence rates with intervention, adverse event rates, proportion of completed study questionnaires, accelerometry and proportion of complete data extraction from ATOMIC app
Utility of the ATOMIC program | Interview [30 minutes] at baseline
  Utility will be addressed through semi-structured interviews that includes both open and closed ended questions. The interviews will be used to elicit the perceptions and preferences of the participants surrounding the use and method of delivery of the PA coaching and program content (e.g. phone, text messaging, posts to app); the usefulness, relevance, and applicability of the ATOMIC program content; as well as facilitators and barriers to use of the program. Semi-structured interviews will be conducted at baseline, six weeks, and post-intervention (twelve weeks). To supplement the interview data, utility will also be captured by counting the number of log-ins to the app and the number of completed coaching sessions and modules.
Utility of the ATOMIC program | Interview [30 minutes] at 6 weeks
  Utility will be addressed through semi-structured interviews that includes both open and closed ended questions. The interviews will be used to elicit the perceptions and preferences of the participants surrounding the use and method of delivery of the PA coaching and program content (e.g. phone, text messaging, posts to app); the usefulness, relevance, and applicability of the ATOMIC program content; as well as facilitators and barriers to use of the program. Semi-structured interviews will be conducted at baseline, six weeks, and post-intervention (twelve weeks). To supplement the interview data, utility will also be captured by counting the number of log-ins to the app and the number of completed coaching sessions and modules.
Utility of the ATOMIC program | Interview [30 minutes] at 12 weeks
  Utility will be addressed through semi-structured interviews that includes both open and closed ended questions. The interviews will be used to elicit the perceptions and preferences of the participants surrounding the use and method of delivery of the PA coaching and program content (e.g. phone, text messaging, posts to app); the usefulness, relevance, and applicability of the ATOMIC program content; as well as facilitators and barriers to use of the program. Semi-structured interviews will be conducted at baseline, six weeks, and post-intervention (twelve weeks). To supplement the interview data, utility will also be captured by counting the number of log-ins to the app and the number of completed coaching sessions and modules.

OTHER OUTCOMES:
Effect of our physical activity (PA) intervention on MVPA level and the mediators of SCT | Entire study - Social Cognitive Mediators and Moderators of Physical Activity scales are completed at baseline, 6 weeks, 12 weeks, and 24 weeks.
  The effect of our PA intervention on MVPA level and the mediators and moderators of SCT (e.g. self efficacy) will be determined by calculating the change in time spent in MVPA and mediators and moderators of SCT at the completion of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No